CLINICAL TRIAL: NCT03045796
Title: Cardiac Output and Central-Venous Oxygen Saturation in Maintenance Hemodialysis Patients
Brief Title: Hypoxemia in Maintenance Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Renal Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 17117
Record Dates: First submitted 2016-11-14; First posted 2017-02-08 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2016-11

CONDITIONS: Oxygen Saturation and the Relationship to Other Cardiac Variables; Maintenance Hemodialysis; Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Maintenance Hemodialysis Patients: Following the initial recruitment, all individuals who are willing to participate and sign the informed consent document will be provided with a medical history form to complete. In addition, we will ask them to sign a HIPAA authorization form in order to look into their medical records for monthly blood work (blood chemistry), anthropometric data (height and weight), interdialytic weight gain (weight gain since last treatment) history, and current medications.
  Interventions: Device: Oxygen Saturation measured by WristOx

INTERVENTIONS:
Device: Oxygen Saturation measured by WristOx — Patients will be hooked up to finger cuffs as well as ECGs to monitor oxygen saturations in different part of the body.

SUMMARY:
Previous research has shown that many patients with kidney failure undergoing chronic hemodialysis (HD) have a very low venous oxygen concentration, which may further decrease during dialysis treatments. This may be due to a variety of factors including anemia, compromised pulmonary function, and chronic fluid volume overload. Previous studies have shown that low venous oxygen concentrations may increase the risk of cardiovascular events, cognitive deficits, and mortality in HD patients.

The purpose of this study is to identify patients with hypoxemia during HD treatments and characterize the extent of and implications of their hypoxemia. Specifically, the investigators aim to examine the relationship between central venous oxygen concentration and hemodynamic changes during dialysis treatment. The investigators will evaluate the relationship between cardiac output as measured by the Task Force Monitor and central venous oxygen saturation as measured by the Crit-Line Monitor and Wrist0x2 in HD patient. Data from this study will provide insight into potential mechanisms responsible for side effects associated with dialysis treatment, such as drops in blood pressure and cognitive dysfunction.

DETAILED DESCRIPTION:
Following the initial recruitment, all individuals who are willing to participate and sign the informed consent document will be provided with a medical history form to complete. In addition, the investigators will ask participants to sign a HIPAA authorization form in order to look into their medical records for monthly blood work (blood chemistry), anthropometric data (height and weight), interdialytic weight gain (weight gain since last treatment) history, and current medications.

Testing DURING all study protocol days:

Testing will be performed on three consecutive dialysis days during a one-week period (Monday/ Wednesday/Friday or Tuesday/Thursday/Saturday). If a data collection period is missed for any reason, an alternative data collection day will be scheduled. All three study visits are identical with respect to the study procedures performed:

1. Hemodynamics: The hemodynamic response to dialysis will be obtained using the Task Force Monitor (TFM). The TFM will be connected to the subject prior the start of the HD session. The TFM is a non-invasive device that uses thoracic bioimpedance to collect a variety of data related to cardiovascular function, including:

   Heart Rate Variability: Beat-to-beat heart rate (HR) will be recorded using the Task Force Monitor. The ECG will be collected online at a sampling rate of 1,000 Hz, in real time, and stored on a computer (Dell, Austin, TX). Heart rate and the variability of the intervals between successive heart rates will be derived from the ECG signal.

   Beat-to-Beat Blood Pressure: Beat-to-beat peripheral BP will be derived via finger plethysmography (Task Force Monitor). A finger cuff will be placed around the non-dialyzing index and middle finger. These cuffs measure the change in blood pressure from successive beats continuously.

   Cardiac Output: Cardiac output and stroke volume will be collected by the task force monitor. An electrode will be placed around the chest to measure changes in impedance continuously.

   Blood Pressure: Blood pressure will be measured before the start and every 10 minutes throughout the session using an automated cuff connected to the TFM. The cuff will be placed on the non-dialyzing arm of the patient. The continuous non-invasive arterial pressure (CNAP) technology on the TFM machine will also be performed continuously during 10 minute segments every hour until the end of the HD treatment (i.e. from minute 0 to 10, 60 to 70, 120 to 130, 180 to 190).

   The TFM will measure these hemodynamic values continuously throughout the entire HD session.
2. Relative Blood Volume and Hematocrit: The Critline is a regular part of dialysis treatment at the Champaign Urbana clinic. The Critline non-invasively measures hematocrit, relative blood volume, and oxygen saturation in real time. A trained staff member of the Champaign Urbana Dialysis Clinic will add a disposable blood chamber to the dialysis machine. As blood travels through this chamber hematocrit and oxygen saturation are measured by the absorbance and scattering of light. The hematocrit value is then used to estimate the blood volume relative to the start of the dialysis session.
3. The Wrist0x2 will be connected prior to the HD session and measurements will be recorded continuously throughout the entire HD session.
4. Clinic Factors: The investigators will gather some information collected by the clinic including: participant weight gain since the previous treatment, the volume of fluid removed during the treatment, the composition of the dialysate used during the treatment, and the rate of flow of both the blood and dialysate through the hemodialysis machine during the treatment.
5. Lab Values: The investigators will also obtain results from monthly blood chemistries run on patient's blood samples by the clinic in the month prior to participant enrollment. These values will include but are not limited to information such as serum albumin, phosphorus, and calcium.

After completion of the HD treatment, the patient will be disconnected from the TFM and Wrist0x2.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and able to give written informed consent to the study
2. Central Venous Catheter (CVC) used for vascular access
3. Participants must receive hemodialysis treatment at least 3 days per week.
4. Participants must be on hemodialysis treatment longer than 3 months. Patients on dialysis treatment for < 3 months will be excluded, or have their enrollment postponed, due to physiological changes that typically occur at the onset of dialysis.
5. Participants must have a central-venous catheter as their vascular access site for dialysis, as our aim is to measure venous oxygen concentrations. Patients with A-V fistula's or grafts will be excluded because we are not interested in collecting arterial oxygen concentrations.

Exclusion Criteria:

1. Scheduled renal transplantation during the study
2. Active infection requiring ongoing antibiotics or antivirals
3. Simultaneous participation in another clinical study with potential impact on cardiovascular/hemodynamic parameters

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Maintenance Hemodialysis Patients
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Hemodynamics | 1 week, 3 Hemodialysis Treatments: Patients will be tested during their three regularly schedule hemodialysis treatment sessions in a one week.
  The hemodynamic response to dialysis will be obtained using the Task Force Monitor (TFM). The TFM will be connected to the subject prior the start of the HD session. The TFM is a non-invasive device that uses thoracic bioimpedance to collect a variety of data related to cardiovascular function, including: heart rate variability, beat-to-beat blood pressure, cardiac output, blood pressure.
Relative Blood Volume and Hematocrit | 1 week, 3 Hemodialysis Treatments: Patients will be tested during their three regularly schedule hemodialysis treatment sessions in a one week.
  The Critline is a regular part of dialysis treatment at the Champaign-Urbana clinic. The Critline non-invasively measures hematocrit, relative blood volume, and oxygen saturation in real time. A trained staff member of the Champaign-Urbana Dialysis Clinic will add a disposable blood chamber to the dialysis machine. As blood travels through this chamber hematocrit and oxygen saturation are measured by the absorbance and scattering of light. The hematocrit value is then used to estimate the blood volume relative to the start of the dialysis session.
Oxygen Saturation | 1 week, 3 Hemodialysis Treatments: Patients will be tested during their three regularly schedule hemodialysis treatment sessions in a one week.
  The Wrist0x2 will be connected prior to the HD session and measurements will be recorded continuously throughout the entire HD session.
Lab Values | 1 week, 3 Hemodialysis Treatments: Patients will be tested during their three regularly schedule hemodialysis treatment sessions in a one week.
  We will also obtain results from monthly blood chemistries run on patient's blood samples by the clinic in the month prior to participant enrollment. These values will include but are not limited to information such as serum albumin, phosphorus, and calcium.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States